CLINICAL TRIAL: NCT02653157
Title: IGHID 11519 - Multidrug Resistant Gram-negative Bacilli Colonization and Infection in Burn
Brief Title: Multidrug Resistant Gram-negative Bacilli Colonization and Infection in Burn
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-1505; US NIH Grant KL2TR001109 (Other Grant/Funding Number: US NIH)
Record Dates: First submitted 2015-10-19; First posted 2016-01-12 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Multi-drug Resistant Gram-negative Bacilli Colonization
Keywords: multidrug resistance; burns; infections, gram-negative bacilli; ventilator-associated pneumonia; ventilator-associated tracheobronchitis; gram-negative bacilli colonization
MeSH Terms: conditions — Burns; Infections; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gram-negative bacterial isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Burn patients with VAT or VAP with MDR-GNB: Adult patients with burn and/or inhalation injury requiring intubation
  Interventions: Other: MDR-GNB

INTERVENTIONS:
Other: MDR-GNB

SUMMARY:
This is a prospective observational study to determine the role of colonization and identify the timing of development of drug resistance in multidrug resistant Gram-negative bacilli (MDR-GNB) causing infection among critically ill burn patients.

DETAILED DESCRIPTION:
This is a prospective observational study. Patients will be followed during a single admission for development of colonization or infection with MDR-GNB. Patient clinical characteristics, including infections, surgeries, and antibiotic exposure, will be collected in real-time.

Weekly surveillance wound and peri-rectal swabs and, if intubated, biweekly deep endotracheal or tracheostomy aspirates will be collected, de-identified, and stored from all patients and examined for the presence of MDR-GNB. All GNB isolates from blood, urine, respiratory, and wound cultures will be collected, coded, and stored.

ELIGIBILITY:
Inclusion Criteria:

1. Severe burn injury, including partial or full thickness burn 20% or more total body surface area; or
2. inhalation injury; or
3. 18 years of age or older;

Exclusion Criteria:

1. Intensive care unit stay of less than 5 days;
2. ICU admission more than 48 hours after burn trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) hospitalized in the NC Jaycee Burn Center who require intubation at or less than 24 hours prior to admission as well as those with 20% or more total body surface area burn, with the anticipation that these patients will subsequently require intubation.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Species causing MDR-GNB colonization | From hospital admission through length of hospital stay, or date of death from any cause, whichever comes first (assessed up to 52 weeks)
  Endotracheal tube or tracheostomy aspirates will be obtained upon admission and twice weekly; wound and perirectal area swabs will be collected weekly and will be used to characterize species.
Time to MDR-GNB colonization | From hospital admission until discharge from unit, or date of death from any cause (assessed up to 1 year)
  surveillance samples for bacterial colonization will be collected weekly
Time to development of MDR and extreme drug resistant bacteria | From hospital admission until date of development of MDR or extremely drug resistant bacteria (assessed up to 52 weeks)
  surveillance samples will be collected weekly
Time to VAT/VAP | Time of hospital admission until date of development of VAT/VAP or date of death from any cause (assessed up to 52 weeks)
  defined by bacteria obtained from clinical bronchoscopy and patient symptoms as noted by chart review
Time to MDR-GNB VAT/VAP | From hospital admission until date of development of MDR-GNB VAT/VAP or date of death from any cause (assessed up to 52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lachiewicz, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Jaycee Burn Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Antibiotic resistance threats in the United States, 2013. Available at http://www.cdc.gov/drugresistance/threat-report-2013 Accessed December 23, 2014.
- [Background] Mosier MJ, Pham TN. American Burn Association Practice guidelines for prevention, diagnosis, and treatment of ventilator-associated pneumonia (VAP) in burn patients. J Burn Care Res. 2009 Nov-Dec;30(6):910-28. doi: 10.1097/BCR.0b013e3181bfb68f. PMID 19826271
- [Background] Brusselaers N, Logie D, Vogelaers D, Monstrey S, Blot S. Burns, inhalation injury and ventilator-associated pneumonia: value of routine surveillance cultures. Burns. 2012 May;38(3):364-70. doi: 10.1016/j.burns.2011.09.005. Epub 2011 Oct 29. PMID 22040929
- [Background] Rue LW 3rd, Cioffi WG, Mason AD Jr, McManus WF, Pruitt BA Jr. The risk of pneumonia in thermally injured patients requiring ventilatory support. J Burn Care Rehabil. 1995 May-Jun;16(3 Pt 1):262-8. doi: 10.1097/00004630-199505000-00008. PMID 7673306
- [Background] Shirani KZ, Pruitt BA Jr, Mason AD Jr. The influence of inhalation injury and pneumonia on burn mortality. Ann Surg. 1987 Jan;205(1):82-7. doi: 10.1097/00000658-198701000-00015. PMID 3800465
- [Background] Tedja R, Nowacki A, Fraser T, Fatica C, Griffiths L, Gordon S, Isada C, van Duin D. The impact of multidrug resistance on outcomes in ventilator-associated pneumonia. Am J Infect Control. 2014 May;42(5):542-5. doi: 10.1016/j.ajic.2013.12.009. Epub 2014 Mar 14. PMID 24630700
- [Background] Lachiewicz AM, van Duin D, DiBiase LM, Jones SW, Carson S, Rutala WA, Cairns BA, Weber DJ. Rates of hospital-associated respiratory infections and associated pathogens in a regional burn center, 2008-2012. Infect Control Hosp Epidemiol. 2015 May;36(5):601-3. doi: 10.1017/ice.2014.90. Epub 2015 Jan 28. No abstract available. PMID 25626446
- [Background] Craven DE, Hjalmarson KI. Ventilator-associated tracheobronchitis and pneumonia: thinking outside the box. Clin Infect Dis. 2010 Aug 1;51 Suppl 1:S59-66. doi: 10.1086/653051. PMID 20597674
- [Background] Sievert DM, Ricks P, Edwards JR, Schneider A, Patel J, Srinivasan A, Kallen A, Limbago B, Fridkin S; National Healthcare Safety Network (NHSN) Team and Participating NHSN Facilities. Antimicrobial-resistant pathogens associated with healthcare-associated infections: summary of data reported to the National Healthcare Safety Network at the Centers for Disease Control and Prevention, 2009-2010. Infect Control Hosp Epidemiol. 2013 Jan;34(1):1-14. doi: 10.1086/668770. Epub 2012 Nov 27. PMID 23221186
- [Background] Siegel JD, Rhinehart E, Jackson M, Chiarello L; Healthcare Infection Control Practices Advisory Committee. Management of multidrug-resistant organisms in health care settings, 2006. Am J Infect Control. 2007 Dec;35(10 Suppl 2):S165-93. doi: 10.1016/j.ajic.2007.10.006. No abstract available. PMID 18068814
- [Background] de La Cal MA, Cerda E, Garcia-Hierro P, Lorente L, Sanchez-Concheiro M, Diaz C, van Saene HK. Pneumonia in patients with severe burns : a classification according to the concept of the carrier state. Chest. 2001 Apr;119(4):1160-5. doi: 10.1378/chest.119.4.1160. PMID 11296184
- [Background] American Burn Association. National Burn Repository 2014 Report. Available at http://www.ameriburn.org/2014NBRAnnualReport.pdf. Accessed December 23, 2014.
- [Background] Brusselaers N, Labeau S, Vogelaers D, Blot S. Value of lower respiratory tract surveillance cultures to predict bacterial pathogens in ventilator-associated pneumonia: systematic review and diagnostic test accuracy meta-analysis. Intensive Care Med. 2013 Mar;39(3):365-75. doi: 10.1007/s00134-012-2759-x. Epub 2012 Nov 28. PMID 23188467
- [Background] Weber DJ, van Duin D, DiBiase LM, Hultman CS, Jones SW, Lachiewicz AM, Sickbert-Bennett EE, Brooks RH, Cairns BA, Rutala WA. Healthcare-associated infections among patients in a large burn intensive care unit: incidence and pathogens, 2008-2012. Infect Control Hosp Epidemiol. 2014 Oct;35(10):1304-6. doi: 10.1086/678067. Epub 2014 Sep 2. No abstract available. PMID 25203188
- [Background] Wibbenmeyer L, Danks R, Faucher L, Amelon M, Latenser B, Kealey GP, Herwaldt LA. Prospective analysis of nosocomial infection rates, antibiotic use, and patterns of resistance in a burn population. J Burn Care Res. 2006 Mar-Apr;27(2):152-60. doi: 10.1097/01.BCR.0000203359.32756.F7. PMID 16566558
- [Background] Magiorakos AP, Srinivasan A, Carey RB, Carmeli Y, Falagas ME, Giske CG, Harbarth S, Hindler JF, Kahlmeter G, Olsson-Liljequist B, Paterson DL, Rice LB, Stelling J, Struelens MJ, Vatopoulos A, Weber JT, Monnet DL. Multidrug-resistant, extensively drug-resistant and pandrug-resistant bacteria: an international expert proposal for interim standard definitions for acquired resistance. Clin Microbiol Infect. 2012 Mar;18(3):268-81. doi: 10.1111/j.1469-0691.2011.03570.x. Epub 2011 Jul 27. PMID 21793988
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- See also: University of North Carolina website — http://www.unc.edu